CLINICAL TRIAL: NCT00072917
Title: The Effects of Overfeeding on Obesity-Prone (OP) and Obesity-Resistant (OR) Women
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Daniel H. Bessesen, MD, University of Colorado School of Medicine
Other Study IDs: OVOPOB DK62874 (complted); DK62874
Record Dates: First submitted 2003-11-12; First posted 2003-11-14 (Estimated); Last update posted 2010-01-18 (Estimated); Status verified 2010-01

CONDITIONS: Obesity; Thinness; Weight Gain
Keywords: obesity; thinness; weight gain; physical activity; diet; fat oxidation; hunger; feeding behavior; overfeeding
MeSH Terms: conditions — Obesity; Thinness; Weight Gain; Motor Activity; Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a longitudinal cohort study of how the responses to a 3 day period of controlled overfeeding relate to subsequent weight gain. We hypothesize that thin individuals are resistant to weight gain because they respond to periods of overfeeding by increasing fat oxidation, reducing food intake, and increasing physical activity relative to those who gain weight over time.

ELIGIBILITY:
* Half of the subjects will be women, half will be men,
* age 25-35,
* a range of BMI's from 19-27, for the 'thin subjects' there should be no 1st degree relatives with a BMI>30.
* Subjects should not engage in planned physical activity more than 3 hrs per week.
* For the obesity prone group there should be at least 1 1st degree relative with a BMI>30.

Ages: 25 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects have been recruited through advertisements in local news media and on the internet
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2003-10; Study Completion 2008-06

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Health Sciences Center, Denver, Colorado, United States

REFERENCES:
- [Derived] Rynders CA, Pereira RI, Bergouignan A, Kealey EH, Bessesen DH. Associations Among Dietary Fat Oxidation Responses to Overfeeding and Weight Gain in Obesity-Prone and Resistant Adults. Obesity (Silver Spring). 2018 Nov;26(11):1758-1766. doi: 10.1002/oby.22321. PMID 30358145
- [Derived] Creasy SA, Rynders CA, Bergouignan A, Kealey EH, Bessesen DH. Free-Living Responses in Energy Balance to Short-Term Overfeeding in Adults Differing in Propensity for Obesity. Obesity (Silver Spring). 2018 Apr;26(4):696-702. doi: 10.1002/oby.22121. PMID 29570248